CLINICAL TRIAL: NCT06199089
Title: A Randomized, Double-blind, Placebo-controlled, and Multi-center Clinical Study to Assess Safety and Efficacy of Anti-Human CD38 Monoclonal Antibody CM313 in the Treatment of Primary Immune Thrombocytopenia
Brief Title: A Randomized, Double-blind, Placebo-controlled, and Multi-center Clinical Study of CM313 in the Treatment of Immune Thrombocytopenia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Tianjin People's Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Henan Cancer Hospital (Other Government); Tianjin Medical University Second Hospital (Other); North China University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2023068
Record Dates: First submitted 2023-12-25; First posted 2024-01-10 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (CM313) (Experimental): 30 from 45 enrolled subjects receive CM313: once a week x 8 doses
  Interventions: Drug: CM313 Injection
- Intervention (Placebo) (Placebo Comparator): 15 from 45 enrolled subjects receive placebo: once a week x 8 doses
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: CM313 Injection — Intravenous CM313 administration
  This study adopts a randomized, double-blind, placebo-controlled design method. A total of 45 subjects were randomly assigned to experimental group (CM313, n = 30) and placebo comparator group (Placebo, n = 15) at a ratio of 2:1. Subjects assigned to experimental group were treated with CD38 monoclonal antibody (CM313: 16mg/kg/w) for 8 weeks.
  The first stage is the main research stage (d1-w8), which is the core treatment period. The subjects will receive intravenous infusion of 16mg/kg CM313 once a week for 8 weeks to observe the efficacy and safety during treatment.
  The second stage (w9-w24) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy of CM313 after treatment.
  Arms: Intervention (CM313)
Drug: Placebo Injection — Intravenous Placebo administration
  This study adopts a randomized, double-blind, placebo-controlled design method. A total of 45 subjects were randomly assigned to experimental group (CM313, n = 30) and placebo comparator group (Placebo, n = 15) at a ratio of 2:1. Subjects assigned to placebo comparator group were treated with placebo of CM313 once a week for 8 weeks.
  The first stage is the main research stage (d1-w8), which is the core treatment period. The subjects will receive intravenous infusion of placebo of CM313 once a week for 8 weeks to observe the efficacy and safety during treatment.
  The second stage (w9-w24) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy after placebo administration.
  Arms: Intervention (Placebo)

SUMMARY:
To evaluate the efficacy and safety of CM313 in the treatment of immune thrombocytopenia in patients who have failed glucocorticoid therapy.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for recurrent and refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

The main pathogenesis of ITP is the loss of platelet autoantigen immune tolerance, which leads to abnormal activation of humoral and cellular immunity. It is characterized by antibody mediated platelet destruction and insufficient platelet production by megakaryocytes. The residual long-term autoreactive plasma cells may be a source of therapeutic resistance to autoimmune cytopenia. Antiplatelet specific plasma cells have been detected in the spleen of patients with rituximab refractory ITP. Therefore, the strategy of simply eliminating B cells may not work, because LLPC will continue to produce pathogenic antibodies. However, targeting LLPC becomes a new strategy to treat autoimmune diseases.

CM313, a kind of anti-CD38 antibody, is a new type of monoclonal antibody targeting CD38. It targets plasma cells and has carried out some clinical studies in multiple myeloma, with good therapeutic effects. In addition, the clinical trials of similar CD38 monoclonal antibody drugs, such as daratumumab, in the treatment of autoimmune diseases, including membranous nephropathy, systemic lupus erythematosus (SLE) and ITP, are also being carried out simultaneously. We assume that autologous reaction LLPC may be the cause of treatment failure in some ITP patients. Therefore, the use of CD38 monoclonal antibody to clear long-term surviving plasma cells in ITP patients may be a new strategy for treating ITP patients.

Therefore, the investigators designed this clinical trial to evaluate the efficacy and safety of CM313 in the treatment of immune thrombocytopenia in patients who have failed glucocorticoid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.
* Before enrollment, the subjects have been clinically diagnosed with primary immune thrombocytopenia for no less than three months according to the American Society of Hematology guidelines 2011 Evidence-Based Practice Guideline (Neunert et al. 2011) or the International Consensus Report for the Investigation and Management of Primary Immune Thrombocytopenia (Provan et al. 2010), as applicable locally.
* Patients have failed glucocorticoid therapy (either due to inefficacy, efficacy could not be maintained, or relapse). Patients were required to have a response history (PLT≥50×10^9/L) to standard first-line treatment of ITP (glucocorticoid and/or intravenous immunoglobulin).
* Subjects with a platelet count of <30×10^9/L within the 24 hours prior to the first dose of the study drug; The mean platelet count of at least two separate assessments (at least 1 week apart) <30×10^9/L during the screening visit, and no platelet count > 35×10^9/L.
* ECOG performance status score of ≤2.
* Enrollment of subjects receiving maintenance therapy with a stable dosage is permitted, including glucocorticoids (≤0.5 mg/kg of prednisone or equivalent) or TPO receptor agonists. However, at the time of enrollment, subjects are restricted to using only one concomitant medication with a stable dose, and the concomitant medication must have been stable for a minimum of 4 weeks prior to the initial infusion of the study drug.
* For fertile female patients, a negative pregnancy test result is required. Fertile female and male patients must use effective contraception separately during the study and for 4 or 6 months after the cessation of study drug treatment.
* Subjects comprehensively understand and can adhere to the study protocol requirements and willingly signed the informed consent form.

Exclusion Criteria:

* Subjects with a known allergy to anti-CD38 monoclonal antibodies or excipients, or those who have previously received anti-CD38 monoclonal antibodies with ineffective therapeutic outcomes.
* Subjects who are diagnosed with autoimmune hemolytic anemia or various secondary thrombocytopenic disorders.
* Subjects with history of any thrombotic or embolic events or extensive and severe bleeding, such as hemoptysis, major upper gastrointestinal bleeding, intracranial hemorrhage, or the presence of sepsis or other irregular bleeding within the 12 months preceding the initiation of the first dose of study drug.
* Subjects who have participated in any other investigational drug studies (including vaccine studies) or been exposed to other investigational drugs within the first 4 weeks or 5 half-lives (whichever was longer) prior to the first dose of study drug.
* Subjects who have used anticoagulants or any agents with antiplatelet effects, such as aspirin, within 3 weeks prior to the first dose of study drug.
* Subjects who have received emergency treatment for ITP (e.g., methylprednisolone, platelet transfusion, intravenous immunoglobulin infusion, or thrombopoietin receptor agonist therapy) within 2 weeks prior to the first dose of study drug.
* Subjects who have been treated with medications including azathioprine, danazol, dapsone, cyclosporine A, tacrolimus, and sirolimus within 4 weeks prior to the first dose of study drug. Subjects who have receive anti-CD20 monoclonal antibodies such as rituximab, or medications including cyclophosphamide and vindesine within 6 months prior to the first dose of study drug.
* Subjects who have undergone splenectomy within 6 months prior to the first dose of study drug.
* Subjects who have received live vaccines within 4 weeks prior to the first dose of study drug, or plan to receive any live vaccines during the course of the study.
* Subjects who are diagnosed with Myelodysplastic syndromes (MDS); Subjects with a with a history of malignancy within the 5 years prior to screening (excluding completely cured in situ cervical cancer and non-metastatic skin squamous cell carcinoma or basal cell carcinoma).
* Subjects who have undergone allogeneic stem cell transplantation or organ transplantation.
* Subjects with a clinically significant medical history, as perceived by investigators, that will pose risks to subjects' safety during the study or potentially affect the safety or efficacy analyses, includes major clinical histories such as circulatory system abnormalities, endocrine system abnormalities, nervous system diseases, blood system diseases, immune system diseases, mental diseases and metabolic abnormalities and so on. e.g., subjects with acute myocardial infarction, unstable angina pectoris, or severe arrhythmias (multifocal ventricular premature contractions, ventricular tachycardia, or ventricular fibrillation) within the 6 months before screening ; New York Heart Association (NYHA) class III-IV heart failure; subjects who were known to have had moderate or severe persistent asthma or chronic obstructive pulmonary disease within the 5 years prior to screening, or whose condition was currently poorly controlled;
* Subjects with a history of severe recurrent or chronic infections, or acute infections requiring systemic treatment with antibiotics, antiviral drugs, antiparasitic drugs, anti-amoebic drugs, or antifungal drugs within 4 weeks prior to the first dose and during the screening period, or superficial skin infections requiring systemic treatment within one week prior to the first dose of study drug. Notably, after the resolution of the infection, the subject may be re-screened.
* Subjects with a history of known or suspected immunosuppression, including invasive opportunistic infections such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis pneumonia, and aspergillosis, even if the infection has resolved; or unusually frequent, recurrent, or prolonged infections (as judged by the investigator).
* Significant laboratory abnormalities during screening included:

  1. Alanine aminotransferase or aspartate aminotransferase greater than three times the upper limit of normal (ULN).
  2. Total bilirubin greater than 1.5 times the ULN (note: subjects diagnosed with Gilbert syndrome based on medical records should not be excluded based on this criterion).
  3. absolute neutrophil count < 1500/mm3.
  4. hemoglobin < 9g/dL; IgG < 500 mg/dL.

  f) lymphocyte count < 500/mm3. g) Creatinine clearance (CrCl) < 30 mL/min (i.e., CrCl ≥30 mL/min is allowed)
* Positive for HIV antibodies or syphilis antibodies.
* Subjects test positive for Hepatitis B surface antigen (HBsAg) or subjects test positive for hepatitis B core antibody and HBV-DNA (through polymerase chain reaction testing), or subjects test positive for hepatitis C virus antibody and HCV-RNA during the screening period. Subjects with positive hepatitis B core antibody but negative HBV-DNA can be enrolled, with HBV-DNA monitoring every 4 weeks.
* Pregnant or lactating women, or those intending to conceive or breastfeed during the study; and male partners intending to induce pregnancy during the study.
* Any other conditions unsuitable for participation in this study, as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy after CM313/Placebo treatment at week 8 | 8 weeks
  Proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at week 8 after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period

SECONDARY OUTCOMES:
Evaluation of the efficacy after CM313/Placebo treatment at each visit period | 24 weeks
  Proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least twice the baseline platelet count without bleeding at each visit period after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Evaluation of the complete remission rate after CM313/Placebo treatment at each visit period | 24 weeks
  Proportion of subjects with a platelet count ≥ 100 × 10^9/L without bleeding at each visit period after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Proportion of subjects with a platelet count ≥ 50 × 10^9/L at each visit period | 24 weeks
  Proportion of subjects with a platelet count ≥ 50 × 10^9/L at each visit period in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Time to response (TTR) | 24 weeks
  Time needed from treatment initiation to platelet count ≥30×10^9/L and at least twice the baseline platelet count
Cumulative weeks of platelet ≥30×10^9/L | 24 weeks
  Cumulative weeks of platelet ≥30×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
Cumulative weeks of platelet ≥50×10^9/L | 24 weeks
  Cumulative weeks of platelet ≥50×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
Emergency treatment | 24 weeks
  Percentage of patients who need emergency treatment after CM313/Placebo treatment
Concomitant maintenance drug | 12 weeks
  Changes in concomitant maintenance therapy at week 12 compared with that before CM313/Placebo treatment
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 12 weeks
  Changes of the subjects' numbers in WHO bleeding score after CM313/Placebo treatment according to the reported World Health Organization's Bleeding Scale at week 12. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Adverse events assessment | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after CM313/Placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI

REFERENCES:
- [Derived] Chen Y, Xu Y, Dai J, Sun T, Li H, Hua Z, Zhou Z, Zhou H, Yan Z, Zhao X, Xue F, Liu W, Liu X, Fu R, Wang W, Chi Y, Dong H, Ju M, Dai X, Gu W, Pei X, Yang R, Zhang L. Anti-CD38 monoclonal antibody CM313 for primary immune thrombocytopenia: multicentre, randomised, placebo controlled, phase 2 trial. BMJ. 2025 Oct 21;391:e084314. doi: 10.1136/bmj-2025-084314. PMID 41120215